CLINICAL TRIAL: NCT01324232
Title: A Phase 2, Double-blind, Randomized, Placebo-controlled, Four-arm, Multicenter, Dose-finding Study to Assess the Safety and Efficacy of Three Dose Levels of AVP-923 (Dextromethorphan/Quinidine) in the Treatment of Central Neuropathic Pain in Patients With Multiple Sclerosis
Brief Title: Safety and Efficacy of AVP-923 in the Treatment of Central Neuropathic Pain in Multiple Sclerosis
Acronym: PRIME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avanir Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-AVR-130
Record Dates: First submitted 2011-03-23; First posted 2011-03-28 (Estimated); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-10

CONDITIONS: Central Neuropathic Pain; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — dextromethorphan - quinidine combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- AVP-923-45 (Experimental)
  Interventions: Drug: AVP-923-45
- AVP-923-30 (Experimental)
  Interventions: Drug: AVP-923-30
- AVP-923-20 (Experimental)
  Interventions: Drug: AVP-923-20

INTERVENTIONS:
Drug: AVP-923-45 — AVP-923-45 (dextromethorphan 45 mg/quinidine 10 mg) capsules administered once daily for first 7 days followed by twice daily for 11 weeks of the study to complete 12 weeks of treatment.
  Arms: AVP-923-45
Drug: AVP-923-30 — AVP-923-30 (dextromethorphan 30 mg/quinidine 10 mg) capsules administered once daily for first 7 days followed by twice daily for 11 weeks of the study to complete 12 weeks of treatment.
  Arms: AVP-923-30
Drug: AVP-923-20 — AVP-923-20 (dextromethorphan 20 mg/quinidine 10 mg) capsules administered once daily for first 7 days followed by twice daily for 11 weeks of the study to complete 12 weeks of treatment.
  Other Names: Nuedexta
  Arms: AVP-923-20
Drug: Placebo — Matching placebo capsules administered once daily for first 7 days followed by twice daily for 11 weeks of the study to complete 12 weeks of treatment.
  Arms: Placebo

SUMMARY:
The objectives of the study are to evaluate the safety, tolerability, and efficacy of 3 doses of AVP-923 capsules in the treatment of central neuropathic pain in participants with multiple sclerosis.

DETAILED DESCRIPTION:
The objectives of the study are to evaluate the safety, tolerability, and efficacy of 3 doses of AVP-923 (dextromethorphan [DM]/quinidine [Q]) capsules containing either 45 mg DM and 10 mg Q (AVP-923-45) or 30 mg DM and 10 mg Q (AVP-923-30) or 20 mg DM and 10 mg Q (AVP-923-20) compared to placebo, for the treatment of central neuropathic pain in a population of participants with multiple sclerosis (MS) over a 12-week period. The MS participant population enrolled includes participants with relapsing-remitting multiple sclerosis (RRMS) and participants with secondary progressive multiple sclerosis (SPMS).

ELIGIBILITY:
Main Inclusion Criteria:

Multiple Sclerosis (relapsing-remitting multiple sclerosis [RRMS] or secondary progressive multiple sclerosis [SPMS]), Clinical history and symptoms of central neuropathic pain (dysesthetic pain) for at least 3 months prior to screening, pain rating scale (PRS) baseline score = or > 4, No MS relapse within previous 30 days.

Main Exclusion Criteria:

Personal history of complete heart block, QT interval corrected for heart rate (QTc) prolongation, or torsades de pointes, family history of congenital QT interval prolongation syndrome, Myasthenia Gravis, Beck Depression Inventory Second Edition (BDI-II) score > 19

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2011-09-08 (Actual); Primary Completion 2013-09-26 (Actual); Study Completion 2013-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (72):
- United States (44):
  - North Central Neurology Associates PC, Cullman, Alabama
  - St. Joseph's Hospital Medical Center, Phoenix, Arizona
  - Alta Bates Summit Medical Center, Berkeley, California
  - University of California, Irvine, Orange, California
  - Coordinated Clinical Research, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Neurology Associates, PA, Maitland, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Laszlo J. Mate, MD, North Palm Beach, Florida
  - Neurology Associates of Ormond Beach, Ormond Beach, Florida
  - Neurological Associates, Pompano Beach, Florida
  - Neurologique Foundation, Ponte Vedra Beach, Florida
  - Suncoast Neuroscience Associates, Inc., St. Petersburg, Florida
  - University of South Florida, Tampa, Florida
  - Geodyssey Research, LLC, Vero Beach, Florida
  - Shepard Center, Atlanta, Georgia
  - Rush-Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Consultants in Neurology, Northbrook, Illinois
  - Josephson Wallack Munshower Neurology, P.C., Indianapolis, Indiana
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan Neurology Associates, P.C., Clinton Township, Michigan
  - Wayne State University, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Advanced Neurology Specialists, Great Falls, Montana
  - Neurology Associates PC, Lincoln, Nebraska
  - Albany Medical Center Hospital, Albany, New York
  - NYU-Hospital for Joint Diseases, New York, New York
  - University of Rochester, Rochester, New York
  - SUNY at Stony Brook, Stony Brook, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Geisinger Health System, Wilkes-Barre, Pennsylvania
  - Advanced Neurosciences Institute, Franklin, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Rocky Mountain MS Clinic, Salt Lake City, Utah
  - Neurological Associates, Henrico, Virginia
  - MS Center of Greater Washington, Vienna, Virginia
  - Swedish Medical Center, Seattle, Washington
  - MultiCare Health System, Tacoma, Washington
- Argentina (8):
  - Instituto de Neurologia Cognitiva, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Hospital Italiano, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto Argentino de Investigacion Neurologica, Ciudad de Buenos Aires, Buenos Aires
  - Hospital Churruca-Visca, Buenos Aires
  - Fundación Argentina Contra las Enfermedades Neurológicas del Envejecimiento - FACENE, Buenos Aires
  - Medeos - Centro de Medicina Integral e Investigación Clínica, Buenos Aires
  - Instituto de Neurología y Neurorrehabilitación del Litoral, Santa Fe
- Czechia (5):
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Jihlava, prispevkova organizace, Jihlava
  - Fakultni Nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
- Poland (9):
  - Szpital Powiatowy w Czeladzi, Czeladź
  - Pomorskie Centrum Traumatologii im. M. Kopernika w Gdansku, Gdansk
  - Zespol Opieki Zdrowotnej w Konskich, Gmina Końskie
  - Diagnomed Clinical Research Sp. z.o.o., Katowice
  - Niepubliczny Zaklad Opieki Zdrowotnej NEURO-MEDIC, Katowice
  - Niepubliczny Zaklad Opieki Zdrowotnej PROFILAKTYKA, Katowice
  - Specjalistyczny Gabinet Neurologiczny, Plewiska
  - Niepubliczny Zaklad Opieki Zdrowotnej NEURO-KARD Ilkowski i Partnerzy Spolka Partnerska Lekarzy, Poznan
  - Osrodek Badan Klinicznych Indywidualnej Specjalistycznej Praktyki Lekarskiej, Szczecin
- Spain (6):
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Vall D´Hebron, Barcelona, Catalonia
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona, Catalonia
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Univ. Nuestra Sra. De La Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Vírgen Macarena, Seville

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After screening procedures, participants underwent a 1-week washout period for all analgesic medications, with the exception of ibuprofen in doses that did not exceed 800 milligrams per day (mg/day).
Groups:
- Placebo: Participants received one matching placebo capsule in the morning during the first 7 days of the study. Participants then received one matching placebo capsule twice daily (approximately every 12 hours) during the remaining 11 weeks of the study to complete 12 weeks of treatment.
- AVP-923-20: Participants received one capsule containing 20 milligrams (mg) dextromethorphan (DM) and 10 mg quinidine (Q) (AVP-923-20) in the morning during the first 7 days of the study. Participants then received one capsule of AVP-923-20 twice daily (approximately every 12 hours) during the remaining 11 weeks of the study to complete 12 weeks of treatment.
- AVP-923-30: Participants received one capsule containing 30 mg DM and 10 mg Q (AVP-923-30) in the morning during the first 7 days of the study. Participants then received one capsule of AVP-923-30 twice daily (approximately every 12 hours) during the remaining 11 weeks of the study to complete 12 weeks of treatment.
- AVP-923-45: Participants received one capsule containing 45 mg DM and 10 mg Q (AVP-923-45) in the morning during the first 7 days of the study. Participants then received one capsule of AVP-923-45 twice daily (approximately every 12 hours) during the remaining 11 weeks of the study to complete 12 weeks of treatment.
Period: Overall Study
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45
Started | 49 | 53 | 54 | 53
Completed | 44 | 42 | 41 | 42
Not Completed | 5 | 11 | 13 | 11
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Missing | 0 | 0 | 1 | 0
Not completed — Participant's Personal Reason/Decision | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 2 | 1 | 2 | 2
Not completed — Participant Refused Medication | 0 | 1 | 0 | 0
Not completed — Intercurrent illness | 0 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 5 | 6 | 6
Not completed — Withdrawal by Subject | 0 | 3 | 4 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45 | Total
Number analyzed (Participants) | 49 | 53 | 54 | 53 | 209
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (8.41) | 47.2 (9.20) | 49.1 (11.21) | 48.1 (13.04) | 48.5 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 12 | 12 | 40
  Male | 40 | 46 | 42 | 41 | 169
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 43 | 46 | 49 | 48 | 186
  Black or African American | 3 | 4 | 5 | 4 | 16
  Asian | 1 | 0 | 0 | 0 | 1
  Hispanic or Latino | 2 | 3 | 0 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Association Between the Dextromethorphan Plasma Concentration and the Change From Baseline Pain Rating Scale (PRS) Score to the Average Pain Rating Scale Score During Days 57 Through 84
Description: PRS required participants to rate their pain over the past 12 hours (hrs) on a scale of 0 to 10 (0=no pain; 10=worst possible pain). Baseline (B) PRS was defined as the average of the PRS scores in the last 7 days collected prior to the B visit. If participants did not have at least 4 PRS scores during the last 7 days prior to the B visit, then the average of up to 7 of the most recent PRS scores available prior to the B visit was used. Post-B PRS was the average of Days 57 through 84 values. For participants who did not have any PRS scores during Days 57 through 84, the average of the last 7 available post-B PRS scores was used. Change from B was calculated as the post-B score minus B score. The average logarithms of dextromethorphan plasma concentrations (Cmax) on Days 22 and 50 are reported in primary outcome measure #2 below. Pearson correlation was calculated between Cmax as one group of data across the reporting groups and Change from Baseline in PRS score.
Time Frame: Baseline; Days 57 through 84 (PRS score); Days 22 and 50 (dextromethorphan plasma concentrations)
Population: Modified Intention-To-Treat (MITT) Population: all participants in the ITT Population (randomized participants) who received at least one dose of study drug, provided a Baseline PRS score, and had at least one post-Baseline PRS assessment. Analysis was based on the randomized treatment assigned (regardless of actual treatment received).
Measure: Median (Full Range); unit: units on a scale
Groups:
- Total: All participants who received placebo, AVP-923-20, AVP-923-30, or AVP-923-45 treatments during the study.
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45 | Total
Number analyzed (Participants) | 49 | 53 | 54 | 53 | 209
units on a scale | -1.821 [-7.86 to 2.06] | -2.143 [-7.60 to 5.71] | -2.650 [-6.54 to 3.00] | -1.679 [-6.79 to 2.00] | -2.000 [-7.86 to 5.71]
Statistical Analysis 1: Comparison: Total; The null hypothesis that the true correlation between the change from Baseline PRS scores and the DM plasma concentration was equal to zero and was tested using a 2-sided test at the 5% level of significance within active treatment groups. The regression line was fitted using change from baseline in average PRS during Day 57-84 as the dependent variable and the average of log-transformed DM Plasma Concentration at Day 22 and Day 50 as the independent variable; Test type: Superiority; p = 0.9827, t-test, 2 sided; Pearson correlation = 0.0019

2. Primary Outcome: Average Logarithms of Dextromethorphan (DM) Plasma Concentrations (Cmax) on Days 22 and 50
Description: The average of the logarithms of the DM plasma concentrations on Days 22 and 50 were presented.
Time Frame: 0 to 3 hours post-dose on Day 22 and 50
Population: MITT Population. Only participants with available data were analyzed.
Measure: Median (Full Range); unit: Log Micrograms per Liter
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45 | Total
Number analyzed (Participants) | 0 | 43 | 45 | 45 | 133
Log Micrograms per Liter |  | 4.019 [2.38 to 4.84] | 4.493 [3.27 to 5.55] | 4.758 [-1.61 to 5.81] | 4.394 [-1.61 to 5.81]

3. Secondary Outcome: Comparison of the Adjusted Mean Change From Baseline PRS Score to the Average PRS Score During Days 57 Through 84
Description: The PRS required participants to rate their pain over the past 12 hours on a scale of 0 to 10 (0=no pain; 10=worst possible pain) by circling the number that best described their pain on average over the past 12 hours. Baseline PRS was defined as the average of the PRS scores in the last 7 days collected prior to the Baseline visit. If participants did not have at least 4 PRS scores during the last 7 days prior to the Baseline visit, then the average of up to 7 of the most recent PRS scores available prior to the Baseline visit was used. Post-Baseline PRS was the average of the Day 57 through 84 values. For participants who did not have any PRS scores during Days 57 through 84, the average of the last 7 available post-Baseline PRS scores was used. Change from Baseline was calculated as the post-Baseline score minus the Baseline score.
Time Frame: Baseline; Days 57 through 84
Population: MITT Population. Analysis was carried out using an analysis of covariance (ANCOVA) model, with the PRS score change from Baseline to Days 57-84 as the dependent variable, treatment group as a fixed effect, and the Baseline PRS score as a covariate.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- AVP-923-20 and AVP-923-30: Participants received either AVP-923-20 or AVP-923-30 in the morning during the first 7 days of the study. Participants then received one capsule of AVP-20 or AVP-923-30 twice daily (approximately every 12 hours) during the remaining 11 weeks of the study to complete 12 weeks of treatment.
- AVP-923-30 and AVP-923-45: Participants received either AVP-923-30 or AVP-923-45 in the morning during the first 7 days of the study. Participants then received one capsule of AVP-923-30 or AVP-923-45 twice daily (approximately every 12 hours) during the remaining 11 weeks of the study to complete 12 weeks of treatment.
- All AVP-923: All participants receiving AVP-923-20, AVP-923-30, or AVP-923-45.
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45 | AVP-923-20 and AVP-923-30 | AVP-923-30 and AVP-923-45 | All AVP-923
Number analyzed (Participants) | 49 | 53 | 54 | 53 | 107 | 107 | 160
units on a scale | -2.04 (0.332) | -2.07 (0.319) | -2.41 (0.316) | -2.00 (0.319) | -2.24 (0.224) | -2.21 (0.225) | -2.16 (0.184)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45 vs AVP-923-20 and AVP-923-30 vs AVP-923-30 and AVP-923-45 vs All AVP-923; Test of dose trend (overall P value); Test type: Superiority; p = 0.8869, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs AVP-923-20; Pairwise treatment group vs placebo; Test type: Superiority; p = 0.9381, ANCOVA; Adjusted mean difference = -0.04, 95% CI 2-sided [-0.94 to 0.87], Standard Error of Mean 0.46
Statistical Analysis 3: Comparison: Placebo vs AVP-923-30; Pairwise treatment group vs placebo; Test type: Superiority; p = 0.4128, ANCOVA; Adjusted mean difference = -0.38, 95% CI 2-sided [-1.28 to 0.53], Standard Error of Mean 0.46
Statistical Analysis 4: Comparison: Placebo vs AVP-923-45; Pairwise treatment group vs placebo; Test type: Superiority; p = 0.9427, ANCOVA; Adjusted mean difference = 0.03, 95% CI 2-sided [-0.88 to 0.94], Standard Error of Mean 0.461
Statistical Analysis 5: Comparison: Placebo vs AVP-923-20 and AVP-923-30; Pairwise treatment group vs placebo; Test type: Superiority; p = 0.6075, ANCOVA; Adjusted mean difference = -0.21, 95% CI 2-sided [-1.0 to 0.58], Standard Error of Mean 0.401
Statistical Analysis 6: Comparison: Placebo vs AVP-923-30 and AVP-923-45; Pairwise treatment group vs placebo; Test type: Superiority; p = 0.6690, ANCOVA; Adjusted mean difference = -0.17, 95% CI 2-sided [-0.96 to 0.62], Standard Error of Mean 0.402
Statistical Analysis 7: Comparison: Placebo vs All AVP-923; Pairwise treatment group vs placebo; Test type: Superiority; p = 0.7394, ANCOVA; Adjusted mean difference = -0.13, 95% CI 2-sided [-0.88 to 0.62], Standard Error of Mean 0.38

4. Secondary Outcome: Mean Change From Baseline in Fatigue Severity Scale (FSS) Scores at Days 57 Through 84
Description: The FSS questionnaire consisted of 9 statements that attempted to explore the severity of fatigue symptoms in participants with MS and other conditions, including chronic fatigue immune dysfunction syndrome and systemic lupus erythematosus, and was designed to differentiate fatigue from clinical depression because both share some of the same symptoms. Participants were asked to respond to each statement on a scale of 1 to 7, with 1 indicating "Strongly Disagree" and 7 indicating "Strongly Agree." Total score ranging from 9 to 63, was computed as the sum of the sub-scores for all 9 statements; a higher score indicated increasing fatigue. Baseline was defined as last non-missing measurement prior to dosing. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Post-Baseline FSS score was the average of Day 57 through 84 values. The analysis was carried out using an ANCOVA model, with the FSS change from Baseline to Days 85 as the dependent variable,
Time Frame: Baseline; Days 57 through 84
Population: MITT Population. Only those participants with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45
Number analyzed (Participants) | 48 | 52 | 54 | 53
units on a scale | -3.32 (1.742) | -2.00 (1.680) | -6.32 (1.642) | -2.12 (1.662)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; Test type: Superiority; p = 0.9731, ANCOVA — The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect
Statistical Analysis 2: Comparison: Placebo vs AVP-923-20; Test type: Superiority; Mean difference (final values) = 1.32, 95% CI 2-sided [-3.46 to 6.09], Standard Error of Mean 2.42
Statistical Analysis 3: Comparison: Placebo vs AVP-923-30; Test type: Superiority; Mean difference (final values) = -3, 95% CI 2-sided [-7.72 to 1.72], Standard Error of Mean 2.394
Statistical Analysis 4: Comparison: Placebo vs AVP-923-45; Test type: Superiority; Mean difference (final values) = 1.2, 95% CI 2-sided [-3.54 to 5.95], Standard Error of Mean 2.408

5. Secondary Outcome: Mean Change From Baseline in Expanded Disability Status Scale (EDSS) Scores at Days 22 and 85
Description: The EDSS, a method of quantifying disability in participants with MS was based on neurological examination of 8 functional systems (FS) (pyramidal, cerebellar, brainstem, sensory, bowel and bladder, visual, cerebral, and other) that allowed neurologists to assign a FS score to each of these systems. Neurological findings in each FS were scored on a scale of 0 (low level of problems) to 5 (high level of problems). The "other" category was not rated numerically but measured disability related to a particular issue, like motor loss. A total averaged EDSS score was then calculated on a scale of 0 (normal) to 10 (death from MS). The total EDSS score was determined by 2 factors: gait and FS scores. A higher score indicated greater disability. Baseline was defined as last non-missing measurement prior to dosing. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline; Days 22 and 85
Population: Safety Population: all participants who received at least 1 dose of study drug. Only participants with a value at both the Baseline visit and the specific post-Baseline visit have been included in the analysis. Safety analyses were performed on the safety population based on the treatment participants actually received.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Total: All participants receiving placebo, AVP-923-20, AVP-923-30, or AVP-923-45.
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45 | Total
Number analyzed (Participants) | 49 | 54 | 53 | 53 | 209
units on a scale
  Day 22: number analyzed (Participants) | 46 | 41 | 42 | 45 | 174
  Day 22 | -0.1 (0.35) | -0.1 (0.56) | -0.2 (0.67) | -0.0 (0.63) | -0.1 (0.56)
  Day 85: number analyzed (Participants) | 48 | 51 | 49 | 52 | 200
  Day 85 | -0.1 (0.75) | -0.1 (0.67) | -0.1 (0.46) | 0.0 (0.58) | -0.1 (0.62)

6. Secondary Outcome: Mean Change From Baseline in Multiple Sclerosis Impact Scale-29 (MSIS-29) Scores at Day 85
Description: MSIS-29, an instrument measuring the physical (20 items) and psychological (9 items) impact of MS from the participants' perspective was used to evaluate therapeutic effectiveness from the participants' perspective. Participants were asked to circle the response that best described the impact of MS on daily life on a scale of 0 (not at all) to 5 (extremely). The total MSIS-29 score ranged from 0 to 145, was calculated as the sum of the sub-scores for all 29 questions, with lower scores indicating better quality of life. Baseline was defined as last non-missing measurement prior to dosing. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was carried out using an ANCOVA model, with the MSIS-29 score change from Baseline to Day 85 as the dependent variable, treatment group as a fixed effect, and the Baseline MSIS-29 as a covariate.
Time Frame: Baseline; Day 85
Population: MITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45
Number analyzed (Participants) | 49 | 53 | 54 | 53
units on a scale | -4.84 (2.651) | -4.34 (2.551) | -6.50 (2.526) | -1.41 (2.550)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect; Test type: Superiority; p = 0.4778, ANCOVA — The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect
Statistical Analysis 2: Comparison: Placebo vs AVP-923-20; Test type: Superiority; Adjusted mean difference = 0.49, 95% CI 2-sided [-6.76 to 7.74], Standard Error of Mean 3.676
Statistical Analysis 3: Comparison: Placebo vs AVP-923-30; Test type: Superiority; Adjusted mean difference = -1.67, 95% CI 2-sided [-8.89 to 5.56], Standard Error of Mean 3.663
Statistical Analysis 4: Comparison: Placebo vs AVP-923-45; Test type: Superiority; Adjusted mean difference = 3.43, 95% CI 2-sided [-3.83 to 10.68], Standard Error of Mean 3.681

7. Secondary Outcome: Mean Change From Baseline in Pittsburgh Sleep Quality Index (PSQI) Scores at Day 85
Description: PSQI, a self-rated questionnaire was used to assess sleep quality and disturbances over a 1-month time interval. A total of 19 individual items generated 7 component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component was scored from 0 (no difficulty) to 3 (severe difficulty). The sum of the scores for the 7 components yielded 1 global score (ranging from 0 to 21). Higher PSQI score indicated worse quality of sleep. Baseline was defined as last non-missing measurement prior to dosing. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was carried out using an ANCOVA model, with the PSQI change from Baseline to Day 85 as the dependent variable, treatment group as a fixed effect, and the Baseline PQIS as a covariate.
Time Frame: Baseline; Day 85
Population: MITT Population. For participants with missing data at Day 85, the last available value has been used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45
Number analyzed (Participants) | 49 | 53 | 54 | 53
units on a scale | -0.51 (0.490) | -1.02 (0.471) | -1.36 (0.467) | -1.71 (0.472)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; Test type: Superiority; p = 0.0685, ANCOVA — The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect
Statistical Analysis 2: Comparison: Placebo vs AVP-923-20; Test type: Superiority; Mean difference (final values) = -0.51, 95% CI 2-sided [-1.85 to 0.83], Standard Error of Mean 0.68
Statistical Analysis 3: Comparison: Placebo vs AVP-923-30; Test type: Superiority; Mean difference (final values) = -0.85, 95% CI 2-sided [-2.19 to 0.48], Standard Error of Mean 0.677
Statistical Analysis 4: Comparison: Placebo vs AVP-923-45; Test type: Superiority; Mean difference (final values) = -1.2, 95% CI 2-sided [-2.54 to 0.15], Standard Error of Mean 0.681

8. Secondary Outcome: Mean Change From Baseline in MS Neuropsychological Screening Questionnaire (MSNQ) Scores at Day 85
Description: MSNQ, a self-reporting, 15-item questionnaire was used to screen for cognitive impairment in participants with MS. Participants (or their informants) scored each item on a scale from 0 (not at all) to 4 (often and greatly interferes with life). The total MSNQ score was calculated as the sum of the sub-scores for all 15 questions and thus ranged from 0 to 60. A higher score indicated greater impairment. Baseline was defined as last non-missing measurement prior to dosing. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was carried out using an ANCOVA model, with the MSNQ score change from Baseline to Day 85 as the dependent variable, treatment group as a fixed effect, and the Baseline MSNQ as a covariate.
Time Frame: Baseline; Day 85
Population: MITT Population. Only those participants with available data were analyzed. For participants with missing data at Day 85, the last available value has been used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45
Number analyzed (Participants) | 48 | 52 | 54 | 53
units on a scale | -0.99 (1.058) | -1.48 (1.020) | -1.88 (0.998) | 0.47 (1.006)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; Test type: Superiority; p = 0.4201, ANCOVA — The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect
Statistical Analysis 2: Comparison: Placebo vs AVP-923-20; Test type: Superiority; Adjusted mean difference = -0.49, 95% CI 2-sided [-3.40 to 2.41], Standard Error of Mean 1.473
Statistical Analysis 3: Comparison: Placebo vs AVP-923-30; Test type: Superiority; Adjusted mean difference = -0.90, 95% CI 2-sided [-3.76 to 1.97], Standard Error of Mean 1.454
Statistical Analysis 4: Comparison: Placebo vs AVP-923-45; Test type: Superiority; Adjusted mean difference = 1.46, 95% CI 2-sided [-1.42 to 4.34], Standard Error of Mean 1.46

9. Secondary Outcome: Mean Change From Baseline in Beck Depression Inventory (BDI-II) Scores at Day 85
Description: BDI-II, a 21-item, self-reported instrument was used to assess the existence and severity of symptoms of depression. Each item corresponded to a symptom of depression and as scored on a 4-point scale, ranging from 0 to 3. Participants were asked to consider each statement as it related to the way they have felt for the past 2 weeks. Each of the 21 items were summed to give a single score for the BDI-II (ranging from 0 to 63). A total score of 0 to 13 indicated minimal depression, a score of 14 to 19 indicated mild depression, a score of 20 to 28 indicated moderate depression, and a score of 29 to 63 indicated severe depression. Baseline was defined as last non-missing measurement prior to dosing. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was carried out using an ANCOVA model, with the BDI-II change from Baseline to Day 85 as the dependent variable, treatment group as a fixed effect, and the Baseline BDI-II as a covariate.
Time Frame: Baseline; Day 85
Population: MITT Population. For participants with missing data at Day 85, the last available value has been used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45
Number analyzed (Participants) | 49 | 53 | 54 | 53
units on a scale | 0.83 (0.868) | -0.26 (0.835) | 0.21 (0.828) | 1.15 (0.837)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect; Test type: Superiority; p = 0.8068, ANCOVA — The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect
Statistical Analysis 2: Comparison: Placebo vs AVP-923-20; Test type: Superiority; Adjusted mean difference = -1.10, 95% CI 2-sided [-3.47 to 1.28], Standard Error of Mean 1.205
Statistical Analysis 3: Comparison: Placebo vs AVP-923-30; Test type: Superiority; Adjusted mean difference = -0.63, 95% CI 2-sided [-2.99 to 1.74], Standard Error of Mean 1.2
Statistical Analysis 4: Comparison: Placebo vs AVP-923-45; Test type: Superiority; Adjusted mean difference = 0.31, 95% CI 2-sided [-2.07 to 2.69], Standard Error of Mean 1.207

10. Secondary Outcome: Mean Change From Baseline in Symbol Digit Modalities Test (SDMT) Scores at Day 85
Description: The SDMT assessed organic cerebral dysfunction in both children (8 years and older) and adults. The SDMT involved a simple substitution task that normal participants could easily perform. Using a reference key, the examinee had 90 seconds to pair specific numbers with given geometric figures. The SDMT score was the total correct response (not counting errors) in 90 seconds and ranged from 0 to 110. Lower scores indicated increased dysfunction. Baseline was defined as last non-missing measurement prior to dosing. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. The analysis was carried out using an ANCOVA model, with the SDMT change from Baseline to Day 85 as the dependent variable, treatment group as a fixed effect, and the Baseline SDMT as a covariate.
Time Frame: Baseline; Day 85
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45
Number analyzed (Participants) | 48 | 52 | 54 | 53
units on a scale
  Total correct responses, Oral: number analyzed (Participants) | 11 | 13 | 20 | 14
  Total correct responses, Oral | 0.59 (2.045) | 2.96 (1.881) | 1.91 (1.525) | 2.06 (1.809)
  Total correct responses, Written: number analyzed (Participants) | 37 | 39 | 34 | 39
  Total correct responses, Written | 1.85 (1.111) | 3.62 (1.086) | 0.16 (1.158) | 0.20 (1.083)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; Test type: Superiority; p = 0.6315, ANCOVA — The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect. Oral responses
Statistical Analysis 2: Comparison: Placebo vs AVP-923-20; Test type: Superiority; Adjusted mean difference = 2.37, 95% CI 2-sided [-3.19 to 7.93], Standard Error of Mean 2.772
Statistical Analysis 3: Comparison: Placebo vs AVP-923-30; Test type: Superiority; Adjusted mean difference = 1.31, 95% CI 2-sided [-3.83 to 6.45], Standard Error of Mean 2.562
Statistical Analysis 4: Comparison: Placebo vs AVP-923-45; Test type: Superiority; Adjusted mean difference = 1.46, 95% CI 2-sided [-4.01 to 6.94], Standard Error of Mean 2.728
Statistical Analysis 5: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; Test type: Superiority; p = 0.1485, ANCOVA — P-value presented tests the hypothesis for overall treatment effect versus no treatment effect. Written responses
Statistical Analysis 6: Comparison: Placebo vs AVP-923-20; Test type: Superiority; Mean difference (final values) = 1.77, 95% CI 2-sided [-1.31 to 4.85], Standard Error of Mean 1.558
Statistical Analysis 7: Comparison: Placebo vs AVP-923-30; Test type: Superiority; Mean difference (final values) = -1.68, 95% CI 2-sided [-4.86 to 1.49], Standard Error of Mean 1.605
Statistical Analysis 8: Comparison: Placebo vs AVP-923-45; Test type: Superiority; Mean difference (final values) = -1.65, 95% CI 2-sided [-4.71 to 1.41], Standard Error of Mean 1.549

11. Secondary Outcome: Mean Numerical Rating Scale (NRS) Scores at Days 22, 50, and 85
Description: The NRS was an 11-point scale for participant self-reporting of pain. The overall scores ranged from 0 (no spasticity) to 10 (worst possible spasticity). Higher scores indicated increased aggression.
Time Frame: Days 22, 50, and 85
Population: MITT Population. Only participants with a value at both the Baseline visit and the specific post-Baseline visit have been included in the analysis. For participants with missing data at Day 85, the last available value has been used.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45 | Total
Number analyzed (Participants) | 49 | 53 | 54 | 53 | 209
units on a scale
  Day 22: number analyzed (Participants) | 42 | 39 | 37 | 40 | 158
  Day 22 | 3.29 (2.717) | 3.56 (3.016) | 3.41 (2.723) | 3.90 (2.649) | 3.54 (2.762)
  Day 50: number analyzed (Participants) | 42 | 37 | 36 | 37 | 152
  Day 50 | 3.24 (2.721) | 2.89 (2.633) | 4.06 (2.888) | 3.54 (2.364) | 3.42 (2.666)
  Day 85: number analyzed (Participants) | 44 | 48 | 46 | 47 | 185
  Day 85 | 3.66 (2.869) | 3.13 (3.085) | 3.87 (2.825) | 3.36 (2.666) | 3.50 (2.857)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; The null hypothesis is that the true correlation between NRS scores and DM plasma concentration is equal to zero. Only 158 of the 209 participants in the mITT Population were analyzed at Day 22; Test type: Superiority; p = 0.1404, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; The null hypothesis that the true correlation between NRS scores and DM plasma concentration is equal to zero. Only 152 of the 209 participants in the mITT Population were analyzed at Day 50; Test type: Superiority; p = 0.0805, t-test, 2 sided
Statistical Analysis 3: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; The null hypothesis that the true correlation between NRS scores and DM plasma concentration is equal to zero. Only 185 of the 209 participants in the mITT Population were analyzed at Day 85; Test type: Superiority; p = 0.0551, t-test, 2 sided

12. Secondary Outcome: Mean Overall Patient Global Impression of Change (PGIC) Scores at Day 85
Description: The PGIC was a standard, validated 7-point categorical scale. The participant was asked to assess the overall change in his or her central neuropathic pain symptoms since entry into the study on a scale of 0 to 7 (0=much better; 7=much worse). Higher scores indicated worsening.
Time Frame: Day 85
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45 | Total
Number analyzed (Participants) | 43 | 45 | 46 | 45 | 179
units on a scale | 3.58 (1.842) | 4.42 (2.398) | 3.70 (2.346) | 3.64 (2.298) | 3.84 (2.244)
Statistical Analysis 1: Comparison: Placebo vs AVP-923-20 vs AVP-923-30 vs AVP-923-45; Test type: Superiority; p = 0.9207, ANCOVA — The p-value presented tests the hypothesis for overall treatment effect versus no treatment effect

13. Other Pre Specified Outcome: Change From Baseline in Modified Ashworth Scale (MAS) Scores
Description: MAS is not considered as a true endpoint. MAS scores were assessed at Baseline only. Change from Baseline could not be calculated because data for the later timepoints was not collected.
Time Frame: Baseline; Day 85
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: AEs were collected up to Week 12.
Description: Treatment-emergent adverse events (AEs) were defined as those events with an onset that was anytime during the study and while on treatment, following the first dose of study drug on Day 1. AEs were reported for members of the Safety Population, comprising all participants who received at least one dose of the study drug. Safety analyses were performed based on the treatment participants actually received.
Arm/Group | Placebo | AVP-923-20 | AVP-923-30 | AVP-923-45
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/54 | 0/53 | 0/53
Serious Adverse Events (participants affected / at risk) | 1/49 | 1/54 | 1/53 | 2/53
Other Adverse Events (participants affected / at risk) | 33/49 | 40/54 | 43/53 | 40/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | AVP-923-20 (N=54) | AVP-923-30 (N=53) | AVP-923-45 (N=53)
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=49) | AVP-923-20 (N=54) | AVP-923-30 (N=53) | AVP-923-45 (N=53)
Dizziness (Nervous system disorders) | 4 | 4 | 9 | 13
Headache (Nervous system disorders) | 6 | 11 | 14 | 8
Multiple sclerosis relapse (Nervous system disorders) | 0 | 2 | 3 | 3
Muscle spasticity (Nervous system disorders) | 2 | 1 | 2 | 3
Neuropathic pain (Nervous system disorders) | 4 | 2 | 3 | 0
Somnolence (Nervous system disorders) | 2 | 5 | 3 | 5
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 2 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 2 | 1
Uhthoff's phenomenon (Nervous system disorders) | 2 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Constipation (Gastrointestinal disorders) | 1 | 3 | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 2 | 3
Nausea (Gastrointestinal disorders) | 7 | 12 | 10 | 8
Vomiting (Gastrointestinal disorders) | 0 | 5 | 2 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Influenza (Infections and infestations) | 0 | 1 | 3 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 2 | 2
Urinary tract infection (Infections and infestations) | 3 | 4 | 5 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 5 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Fatigue (General disorders) | 3 | 3 | 3 | 3
Asthenia (General disorders) | 1 | 2 | 1 | 2
Malaise (General disorders) | 0 | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 1 | 3 | 0
Depression (Psychiatric disorders) | 1 | 0 | 3 | 2
Insomnia (Psychiatric disorders) | 1 | 3 | 2 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 3
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 1 | 5
Ear pain (Ear and labyrinth disorders) | 0 | 2 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 3 | 2
Diplopia (Eye disorders) | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 2 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.